CLINICAL TRIAL: NCT03089827
Title: Biodistribution of [11C]PIB in Patients With Risk Factors for Alzheimer's Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00027675
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Memory
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants enrolled at the Alzheimer's Disease Research Center (ADRC) at Wake Forest School of Medicine will be invited to take part in this study. The purpose of this study is to identify and measure the amount of a protein called amyloid in the brain.It is thought that the build up of amyloid may be related to the development of Alzheimer's disease.

DETAILED DESCRIPTION:
Brain amyloid will be measured using PET with [11C]PiB. Participation will involve an initial brain scan and possibly a follow-up brain scan two years later.

The data collected in this study will help explain amyloid deposits in several groups of participants including adults with and without signs of memory impairment. The information collected will help find out who is more likely to have brain amyloid and when it increases the risk for developing memory problems. Research studies suggest that people with elevated levels of brain amyloid are at an increased risk for memory decline, but this does not mean that every person with amyloid build up will develop AD.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a study with the Alzheimer's Disease Research Center.

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults enrolled with the Alzheimer's Disease Research Center at Wake Forest School of Medicine will be invited to participate,
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-05-21 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Amyloid deposition | 2 years
  Studying the initial amyloid deposition in participants as well as their rate of amyloid accumulation over time will help establish whether there is an early therapeutic window for intervention in high risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No